CLINICAL TRIAL: NCT05377294
Title: Is Method of Levels (MOL) Therapy an Acceptable and Feasible Psychological Intervention for People in Acute Mental Health Inpatient Services: A Case Series.
Brief Title: Acceptability and Feasibility of MOL in Acute Inpatient Units
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Lydia Carr, Ms Lydia Carr, Trainee Clinical Psychologist, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 305321
Record Dates: First submitted 2022-05-08; First posted 2022-05-17 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Psychosis; Suicidal
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MOL therapy (Experimental): Participants with Psychosis and/or Suicidality receiving MOL therapy
  Interventions: Other: Method of Levels therapy

INTERVENTIONS:
Other: Method of Levels therapy — MOL therapy aims to help people develop awareness of their personal goals so they can identify incompatibilities and find potential solutions. In MOL, the therapist uses a specific style to help people focus attention on the problem at hand, long enough to consider the issues from different perspectives, including reflection on the associated emotions. This process is usually very experiential and requires the client to be actively engaged in controlling the focus of the session and decision making.

SUMMARY:
The current study aims to test the acceptability and feasibility of a psychological therapy called Method of Levels (MOL) as an intervention for people in acute psychiatric inpatient units who are experiencing psychosis and/or suicidality.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 18 years
* Current service user in an acute inpatient ward in the Greater Manchester area
* Capacity to provide informed consent for participating in research
* Good command of English language
* WS1: Experiencing psychosis (this will be screened for using a clinical cut-off score on the CAPE (Mossaheb et al., 2012))
* WS2: Experiencing suicidality (this will be screened for using a cynical cut-off score on the Suicidal Behaviours Questionnaire - revised (SBQ-R) (Osman et al., 2001))

Exclusion Criteria:

* Problems of an organic nature or a learning disability that might affect cognitive functioning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Proportion of approved patients recruited | Study consent meeting, approx. 1 week after initial meeting
  We will deem the study feasible if at least 72% of approached people consent to participate
Proportion of recruited patients retained | End of therapy interview
  We will deem the study feasible if least 62% of recruited participants are retained (i.e. receive at least one therapy session and complete the end of therapy measures and interview)
Number of participants who receiving the intervention | End of first therapy session, approx. 2 weeks after initial meeting
  We will deem the study feasible if 10 participants receive at least one therapy session
Acceptability (qualitative) | End of therapy interview
  Qualitative interview with participant at end of therapy analysed using Thematic Analysis
Results of Novel Client Measure (descriptive) | End of therapy research meeting
  Qualitative self-reported perception of what was helpful about the therapeutic environment
Results of Outcome Rating Scale (descriptive) | End of therapy research meeting
  Qualitative self-report measure assessing areas of life functioning known to change as a result of therapeutic intervention
Feasibility of adaptions required | Final follow up meeting with final participant, 3 months after consent
  Qualitative record of adaptions required for use of MOL in an acute inpatient setting

OTHER OUTCOMES:
Psychological Outcomes Profile (descriptive) | End of therapy research meeting
  Outcome measure assessing idiosyncratic problems and distress
Clinical Outcomes in Routine Evaluation-OM (descriptive) | End of therapy research meeting
  Outcome measure assessing idiosyncratic problems and distress
Reorganisation of Conflict Scale (descriptive) | End of therapy research meeting
  Outcome measure assessing goal conflict reorganisation (a key mechanism of change in MOL)
Community Assessment of Psychic Experiences (if experiencing psychosis at point of consent) | End of therapy research meeting
  Outcome measure assessing experiences of psychosis
Linehan Reasons for Living Inventory (if experiencing suicidality at point of consent) | End of therapy research meeting
  Outcome measure assessing experiences of suicidality

CONTACTS AND LOCATIONS:
Overall Officials: Sara Tai, DClinPsy, Principal Investigator — University of Manchester; Yvonne Awenat, PhD, Principal Investigator — University of Manchester
Locations (2):
- United Kingdom (2):
  - GMMH Park House, Manchester
  - GMMH: Laureate House, Manchester

IPD SHARING:
Plan to Share IPD: Undecided